CLINICAL TRIAL: NCT00405444
Title: Intranasal Fentanyl Versus Placebo for Catheterization During a Voiding Cystourethrogram in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Seen Chung/Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000009018
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Pain
Keywords: Pediatrics; Pain; Voiding Cystourethrogram; Catheterization; Fentanyl
MeSH Terms: conditions — Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Fentanyl
- 2 (Placebo Comparator)
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Fentanyl — The dose of fentanyl that each child will receive will be 2 mcg/kg based on the child's weight. The medication will be administered 10 minutes prior to the procedure and will be dropped into the unoccluded nares over 1-2 seconds.
  Arms: 1
Drug: Sterile water — The dose of sterile water that each child will receive will be 2 mcg/kg based on the child's weight. It will be administered 10 minutes prior to the procedure and will be dropped into the unoccluded nares over 1-2 seconds.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether intranasal fentanyl is better than placebo at decreasing pain in children 4-8 years of age during urinary catheterization for a VCUG study.

DETAILED DESCRIPTION:
Studies have shown that the voiding cystourethrogram (VCUG) can be distressful and painful for children as the child is catheterized during the procedure. Currently no sedation or analgesia is recommended for the procedure. The practice of pediatrics is constantly seeking measures to decrease pain and distress for children. The opioid fentanyl was originally synthesized in the 1950's and 60's as an alternative to morphine and meperidine. The safety and efficacy of intranasal (IN) fentanyl has been previously demonstrated in the setting of a pediatric emergency department.

We are proposing the use of IN fentanyl for analgesia prior to the catheterization for a voiding cystourethrogram (VCUG). If we prove that IN fentanyl is effective in reducing the pain while ensuring patient safety, it could become the analgesic of choice for this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4-8 years
2. Scheduled VCUG at Sick Kids
3. Understand the consent and assent form in English

Exclusion Criteria:

1. Previous adverse events to fentanyl or any opioid
2. History of a chronic respiratory or cardiac illness
3. Children with developmental delay
4. Children with bilateral nasal congestion.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in pain before and after catheterization for the VCUG. | Will be measured up until 30 mins after the VCUG procedure.

SECONDARY OUTCOMES:
Heart rate, respiratory rate and oxygen saturation just prior to and after the administration of fentanyl. | Every 5 minutes until 30 minutes after the VCUG procedure.
Nausea, vomiting, itching, nasal pain/irritation or any other side effects. | Will be measured up until 30 mins after the VCUG procedure.
Length of stay in diagnostic suite | Time frame determined by outcome

CONTACTS AND LOCATIONS:
Overall Officials: Seen Chung, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Chung S, Lim R, Goldman RD. Intranasal fentanyl versus placebo for pain in children during catheterization for voiding cystourethrography. Pediatr Radiol. 2010 Jul;40(7):1236-40. doi: 10.1007/s00247-009-1521-1. Epub 2010 Feb 24. PMID 20180109